CLINICAL TRIAL: NCT01677572
Title: A Randomized, Double-Blinded, Placebo-Controlled Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB037 in Subjects With Prodromal or Mild Alzheimer's Disease
Brief Title: Multiple Dose Study of Aducanumab (BIIB037) (Recombinant, Fully Human Anti-Aβ IgG1 mAb) in Participants With Prodromal or Mild Alzheimer's Disease
Acronym: PRIME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was discontinued based on futility analysis conducted on Phase 3 trials (NCT02477800 and NCT02484547) and not based on safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 221AD103; 2012-000349-10 (EudraCT Number)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease
Keywords: Aducanumab; BIIB037
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab; Immunoglobulin G

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Low-dose #1 Aducanumab (Experimental): Intravenous doses of low-dose level #1 Aducanumab administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb)
- Low-dose #2 Aducanumab (Experimental): Intravenous doses of low-dose level #2 Aducanumab administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb)
- Placebo (low dose group) (Placebo Comparator): Intravenous doses of placebo administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb); Drug: Placebo
- Mid-dose Aducanumab (Experimental): Intravenous doses of mid-dose Aducanumab administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb)
- Placebo (mid dose group) (Placebo Comparator): Intravenous doses of placebo administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb); Drug: Placebo
- High-dose Aducanumab (Experimental): Intravenous doses of high-dose Aducanumab administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb)
- Placebo (high dose group) (Placebo Comparator): Intravenous doses of placebo administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose administered approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb); Drug: Placebo
- Aducanumab Titration (Experimental): Intravenous doses of Aducanumab administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb)
- Placebo (Titration Group) (Placebo Comparator): Intravenous doses of placebo administered approximately 4 weeks apart over approximately 52 weeks (a total of 14 doses). Qualifying participants can continue into the long-term extension at a dose approximately 4 weeks apart for up to an additional 112 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb) — Participants will receive an infusion of Aducanumab on Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, and 365 (±2 days) at the study clinic and assigned does levels. The infusion will be administered for approximately 1 hour. The study is conducted with a staggered, parallel group design, with the first 3 treatment arms conducted in parallel, 2 further treatment arms subsequently beginning in parallel and the 2 last treatment arms subsequently beginning in parallel. Qualifying participants can enter the long-term extension period at doses described in the treatment arms for up to an additional 112 doses.
  Other Names: IgG1; anti-A* mAb; Fully human
  Arms: Aducanumab Titration; High-dose Aducanumab; Low-dose #1 Aducanumab; Low-dose #2 Aducanumab; Mid-dose Aducanumab; Placebo (high dose group); Placebo (low dose group); Placebo (mid dose group)
Drug: Placebo — Placebo to mimic the low dose, mid-dose and high-dose treatment arms of the experimental intervention; administered by intravenous (IV) infusion on Days 1, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, and 365 (±2 days) at the study clinic. Qualifying participants can enter the long-term extension period at doses described in the treatment arms for up to an additional 112 doses.
  Arms: Placebo (Titration Group); Placebo (high dose group); Placebo (low dose group); Placebo (mid dose group)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple doses of Aducanumab (recombinant, fully human anti-Aβ IgG1 mAb) in participants with prodromal or mild Alzheimer's Disease (AD). The secondary objectives of this study are to assess the effect on cerebral amyloid plaque content as measured by florbetapir-fluorine-18 (18F-AV-45F-AV-45) positron emission tomography (PET) imaging, to assess the multiple dose serum concentrations of Aducanumab and to evaluate the immunogenicity of Aducanumab after multiple dose administration in this population.

DETAILED DESCRIPTION:
The study consists of a placebo-controlled period to study week 54, followed by a long-term extension to study week 518. The placebo-controlled period is conducted with a staggered, parallel group design, with the first 3 treatment arms conducted in parallel, 2 further treatment arms subsequently beginning in parallel, 2 additional treatment arms beginning in parallel, and the last 2 treatment arms subsequently beginning in parallel. Qualifying participants can enter the long-term extension period for up to 42 additional doses of active drug for the first 3 years of LTE. Furthermore, up until the last participant in Arms 8 and 9 has had his or her last dose in the fifth year of the LTE, eligible participants will be able to continue treatment beyond the third year of the LTE.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be ambulatory.
* Participants must meet the following core clinical criteria as determined by the Investigator:

Prodromal Alzheimer's Disease (AD) (all of the criteria must apply):

* Mini Mental State Examination (MMSE) scores between 24-30 (inclusive)
* a spontaneous memory complaint
* objective memory loss defined as a free recall score of ≤27 on the Free and Cued Selective Reminding Test (FCSRT)
* a global Clinical Dementia Rating Scale (CDR) score of 0.5
* absence of significant levels of impairment in other cognitive domains
* essentially preserved activities of daily living, and an absence of dementia. OR

Mild Alzheimer's Disease (AD) criteria (all criteria must apply):

* Mini Mental State Examination (MMSE) scores between 20-26 (inclusive)
* a global Clinical Dementia Rating Scale (CDR) of 0.5 or 1.0
* meeting the National Institute on Aging-Alzheimer's Association core clinical criteria for probable AD.
* Participants must have a positive florbetapir positron emission tomography (PET) amyloid scan.
* Participants must consent to apolipoprotein E (ApoE) genotyping.
* Apart from clinical diagnosis of Alzheimer's Disease (AD), participant must be in good health.
* Must have a reliable informant or caregiver.

Key Exclusion Criteria:

* Any medical or neurological condition (other than Alzheimer's Disease) that might be a contributing cause of the participant's cognitive impairment.
* Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year.
* Clinically significant psychiatric illness in past 6 months.
* Seizure in the past 3 years.
* Poorly controlled diabetes mellitus.
* History of unstable angina, myocardial infarction, chronic heart failure, or clinical significant conduction abnormalities within 1 year prior to Screening.
* Indication of impaired renal or liver function.
* Have human immunodeficiency virus (HIV) infection.
* Have a significant systematic illness or infection in past 30 days.
* Brain MRI showing evidence of acute or sub-acute micro or macrohemorrhage, greater than 4 microhemorrhages, cortical infarct or greater than one 1 lunar infarct.
* Any contraindications to brain MRI or positron emission tomography (PET) scans.
* Negative positron emission tomography (PET) scan with any amyloid-targeting ligand within 48 weeks of Screening.
* Clinically significant 12-lead electrocardiogram (ECG) abnormalities.
* Alcohol or substance abuse in past 1 year.
* Taking blood thinners (except for aspirin at a prophylactic dose or less)
* Have changes in medications or doses of medication in past 4 weeks.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Baseline to week 518

SECONDARY OUTCOMES:
Change from baseline in florbetapir-fluorine-18 (18F-AV-45F-AV-45) positron emission tomography (PET) imaging in certain brain areas. | Day 1, Weeks 26, 54, End of year 2, 3, and 4
Multiple dose pharmacokinetic (PK) serum concentrations of Aducanumab | Up to week 518
Change from Baseline in Incidence of Anti-Aducanumab Antibodies in Serum. | Up to week 518

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- United States (32):
  - NNS Clinical Research, LLC, Tucson, Arizona
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - University of California, Los Angeles, Los Angeles, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Pacific Research Network, Inc., San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Alzheimer's Disease Research Unit, Yale University, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - MD Clinical Trials, Inc., Hallandale, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Galiz Research, LLC, Miami Springs, Florida
  - Compass Research, LLC, Orlando, Florida
  - Infinity Clinical Research, Inc., Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Neurostudies.net, LLC, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - St. Louis Clinical Trials, LLC, St Louis, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - CRI Lifetree, Marlton, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Empire Neurology, PC, Latham, New York
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Brown Hospital, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Chen T, O'Gorman J, Castrillo-Viguera C, Rajagovindan R, Curiale GG, Tian Y, Patel D, von Rosenstiel P, von Hehn C, Salloway S, Hock C, Nitsch RM, Haeberlein SB, Sandrock A, Singhal P. Results from the long-term extension of PRIME: A randomized Phase 1b trial of aducanumab. Alzheimers Dement. 2024 May;20(5):3406-3415. doi: 10.1002/alz.13755. Epub 2024 Apr 3. PMID 38567735
- [Derived] Sevigny J, Chiao P, Bussiere T, Weinreb PH, Williams L, Maier M, Dunstan R, Salloway S, Chen T, Ling Y, O'Gorman J, Qian F, Arastu M, Li M, Chollate S, Brennan MS, Quintero-Monzon O, Scannevin RH, Arnold HM, Engber T, Rhodes K, Ferrero J, Hang Y, Mikulskis A, Grimm J, Hock C, Nitsch RM, Sandrock A. The antibody aducanumab reduces Abeta plaques in Alzheimer's disease. Nature. 2016 Sep 1;537(7618):50-6. doi: 10.1038/nature19323. PMID 27582220